CLINICAL TRIAL: NCT06884384
Title: Direct Oral Anticoagulants Versus Warfarin in Patients With Non-high-risk Antiphospholipid Syndrome : Prospective Cohort Study
Brief Title: DOAC Versus VKA in Patients With Non-high-risk APS : Prospective Cohort Study
Acronym: DOWAPS
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Virginie Dufrost, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024-A02295-42; 2023-0195 (Other: Promotor code)
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Antiphospholipid Syndrome (APS); Cohort Study; Thrombotic and Bleeding Events
Keywords: Antiphospholipid Syndrome; VKA treatment; DOAC Treatment; biological analysis; Thrombotic and bleeding events
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — all patients will have a blood sample taken at inclusion as part of a routine blood test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with VKA treatment: Population of "non-high-risk" thrombotic APS patients treated with VKAs, regardless of how long they have been on therapy. "Non-high-risk" APS is defined by the absence of a history of arterial or microcirculatory thrombosis, the absence of valvulopathy related to APS and a biological profile with only one or two positive antiphospholipid tests.
  Interventions: Biological: Additional blood collection during routine blood sampling at the inclusion (33.9 ml) and at the thrombotic recurrence (between 3.5 and 5 ml); Behavioral: Completion of a questionnaire on compliance with anticoagulant treatment; Behavioral: Completion of a questionnaire on satisfaction with treatment anticoagulant
- Patient with DOAC treatment: Population of "non-high-risk" thrombotic APS patients treated with oral AntiXa, regardless of how long they have been treated. Non-high-risk" APS is defined by the absence of a history of arterial or microcirculatory thrombosis, the absence of valvulopathy related to APS, and a biological profile with only one or two positive antiphospholipid tests.
  Interventions: Biological: Additional blood collection during routine blood sampling at the inclusion (33.9 ml) and at the thrombotic recurrence (between 3.5 and 5 ml); Behavioral: Completion of a questionnaire on compliance with anticoagulant treatment; Behavioral: Completion of a questionnaire on satisfaction with treatment anticoagulant

INTERVENTIONS:
Biological: Additional blood collection during routine blood sampling at the inclusion (33.9 ml) and at the thrombotic recurrence (between 3.5 and 5 ml) — At inclusion, the blood sample is used to perform thrombin generation tests (activated protein C resistance profile and ratio), classical and innovative aPL assays centrally to limit the fluctuation inherent in the tests used and enable comparison between patients, immunothrombosis markers: circulating neutrophil extracellular traps (NETs) assay, sTREM-1 assay
  In the event of recurrence, blood sampling can be used to confirm compliance with treatment by measuring the anti Xa activity of the drug or INR
Behavioral: Completion of a questionnaire on compliance with anticoagulant treatment — The Girerd questionnaire (6 questions) will be proposed to patients in order to estimate the degree of compliance with AODs and VKAs at inclusion and at each follow-up visit for the duration of their participation in the study.
  Other Names: GIRERD questionnaire
Behavioral: Completion of a questionnaire on satisfaction with treatment anticoagulant — The ACTS questionnaire (15 questions) will be proposed to them in order to estimate their satisfaction with their anticoagulant treatment (AOD or AVK) at inclusion and at each follow-up visit for the duration of their participation in the study.
  Other Names: Anti-Clot Treatment Scale - ACTS

SUMMARY:
Antiphospholipid syndrome (APS) is a thrombotic disease requiring prolonged anticoagulation. Direct oral anticoagulants (DOACs) are indicated as 1st-line therapy in venous thrombosis, compared with VKAs, due to their easier handling and lower bleeding risk for equivalent efficacy. In APS, VKAs are still the reference treatment. However, DOACs are generally introduced in the acute phase of venous, before the diagnosis of APS. VKA have the disadvantage of numerous food and drug interactions, and therefore require close monitoring of INR, at least once a month. Because they are easier to use than VKAs, and the risk of bleeding is lower, patients are often reluctant to switch from DOACs to VKA. Studies have shown that APS patients with high thrombotic risk (positivity of all three antiphospholipid tests, history of arterial or small vessels thrombosis or cardiac valve damage) have an increased thrombotic risk during DOACs vs. VKA treatment. Since 2020, the ISTH guidelines have suggested avoiding DOACs in high-risk APS, but suggest continuing theim in other patients if they were introduced for venous thrombosis and if follow-up on DOACs is reassuring. In the case of high-risk APS patients, the relay is therefore systematic. For non-high-risk patients (the majority), there are no data to justify systematic switch. Given the quality-of-life advantages of DOACs over VKAs, patients are not always in favor of changing their anticoagulant therapy, especially if they have been on it for many years with good tolerability. For these reasons, a number of patients with non-high-risk APS remain on DOACs. Nevertheless, the limited data available on the efficacy of DOACs in non-high-risk patients are of low level of evidence and contradictory. In 2020, a literature review of non-high-risk SAPL patients treated with DOACs reported that 8.6% of them experienced thrombotic recurrence within 12 months, with no possible comparison with VKAs. A recent retrospective study with 96 patients reported that 15.4% of patients treated with DOACs had a recurrence, compared to 5.3% on VKAs. However, this difference was not statistically significant (p=0.15) due to a clear lack of power. The objective is to determine the frequency of thrombotic recurrences and to compare it according to the type of oral treatment, anti-Xa versus VKA, in non-high-risk APS, through a cohort study with prospective follow-up. The patient's usual antithrombotic treatment, DOAC and VKA, will be continued unchanged.

DETAILED DESCRIPTION:
prospective cohort of APS patient treated with VKA or DOACs (specially oral Xa treatment).

APS patients will be non high risk patients (no triple positivity, any previous arterial or small vessels thrombosis or cardiac involvment).

the treatment taken by the patient at inclusion will not be modified. There will therefore be no change to the patient's usual management.

all patients will have a blood sample taken at inclusion as part of a routine blood test.

Patients will be prospectively follow up and the level of recurrence thrombotic event will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Persons who have received full information about the organization of the research and have given their oral consent to participate.
* Male or female 18 years of age or older;
* Carrier of venous thrombotic SAPL:

  * Not favoured by a major or ≥ 2 minor favouring factors, if the patient doesn't present with obstetrical SAPL in accordance with the ACR/EULAR 2023 clinical classification criteria.
  * Or favored by ≥ 2 minors, if the patient has obstetrical SAPL: severe preeclampsia < 34 weeks or placental insufficiency
  * Regardless of how long the disease has been present
  * With persistent positivity of at least one biological criterion:

    * Positivity of circulating lupus anticoagulant or IgG anticardiolipid or IgG anti-beta-2GPI
    * And persistence of the same positive test ≥ 12 weeks apart
    * And With maximum delay of positivity of the 1st antiphospholipid test of 3 years after the thrombotic event
* Current anticoagulant treatment, regardless of date of introduction

  * rivaroxaban or apixaban
  * or antivitamin K
* Patient affiliated to a social security system

Exclusion Criteria:

* Venous thrombotic event motivating current anticoagulant treatment favoured by a major favouring factor:

  * Active cancer
  * Hospitalization with bed rest for at least 3 days in the 3 months preceding the event
  * Major trauma with fractures or spinal cord injury in the month preceding the event
  * Surgery with general/spinal/epidural anesthesia for > 30 minutes in the 3 months preceding the event.
* In the absence of a history of pre-eclampsia or placental insufficiency: venous thrombotic event motivating current anticoagulant treatment favoured by 2 or more minor favouring factors:

  * Systemic autoimmune disease or active inflammatory bowel disease
  * Acute/severe infection
  * Central venous catheter in the same vascular bed
  * Hormone replacement therapy, estrogenic oral contraceptives, or hormone-stimulating therapy in progress
  * Long-distance travel (≥ 8 hours)
  * Obesity (BMI ≥ 30 kg/m²)
  * Pregnancy or post-partum (6 weeks after delivery)
  * Prolonged immobilization
  * Surgery with general/spinal/epidural anesthesia for < 30 minutes in the 3 months preceding the event
* Known triple antiphospholipid positivity
* Isolated IgM antiphospholipid positivity
* History of known arterial thrombosis
* History of known microcirculatory thrombosis
* Known SAPL-related cardiac valvular disease
* Persons referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code
* Persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care under articles L. 3212-1 and L. 3213-1.
* Glomerular filtration rate < 30ml/min.
* Weight < 50kg
* History of thrombotic recurrence under well-administered anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of "non-high-risk" thrombotic APS patients treated with oral AntiXa or VKA regarding the treatment already taken at inclusion. Non-high-risk" APS is defined by no history of arterial or small vessels thrombosis, any valvulopathy related to APS, and a biological profile with only one or two positive antiphospholipid tests.
  Patients will be recruited via the departments authorized to manage them, during their consultation or hospitalization. Patients will be invited to participate in the study as part of their regular follow-up visit. There will be no change in current antithrombotic treatment at the time of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2031-09-15 (Estimated); Study Completion 2031-09-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of thrombotic recurrence between the 2 arms | "From enrollment to the thrombotic recurrence or the end of the study (24 months post-inclusion)
  Occurrence (percentage at group level) of thrombotic recurrence within 24 months of inclusion confirmed by objective examination and defined by the occurrence of one of the following events:
  * Venous thrombosis of any location or pulmonary embolism
  * Arterial thrombosis in any location
  * Microcirculatory thrombosis in any location

SECONDARY OUTCOMES:
Risk Factors of thrombotic recurrence on the 2 arms | Biological parameters : at the end of the study after the last visit of the last patient. No biological parameters : from enrollment to the end of follow-up (24 months post-inclusion or thrombotic recurrence)
  The risk factors for thrombotic recurrence tested were: age, gender, cardiovascular risk factors, manifestations associated with APS, associated autoimmune diseases, biological parameters (antiXa activity, INR, biomarkers of immunothrombosis collected as part of the research.
Occurrence of major hemorrhage between the 2 arms | From enrollment to the end of follow-up (24 month post-inclusion or thrombotic recurrence)
  Major bleeding as defined by the International Society on Thrombosis and Haemostasis within Haemostasis within 24 months of inclusion
Occurrence of clinically relevant hemorrhage between the 2 arms | From enrollment to the end of follow-up (24 months post-inclusion or thrombotic recurrence)
  Occurrence of clinically relevant bleeding as defined by the International Society on Thrombosis and Haemostasis within 24 months of inclusion
Occurrence of a minor bleed between the 2 arms | From enrollment to the end of follow-up (24 months post-inclusion or thrombotic recurrence)
  Occurrence of a minor bleed within 24 months of inclusion, defined as a bleed that does not meet the International Society on Thrombosis and Haemostasis definition of clinically relevant major or non-major bleeding.
Net clinical benefit defined as a composite endpoint between the 2 arms | From enrollment to the end of follow-up (24 months post-inclusion or thrombotic recurrence)
  Net clinical benefit defined as a composite endpoint including venous, arterial or microcirculatory thrombotic recurrence, cardiovascular death or major bleeding as defined by ISTH during 24-month follow-up.
Drug Compliance evaluation between the 2 arms | From enrollment to the end of follow-up (24 months post-inclusion or thrombotic recurrence)
  Drug Compliance score assessed by Girerd test at baseline and follow-up visits. Score between 0 to 6. 0 indicates a good observance, 1 to 2 : minimal observance problem and ≥ 3 : Poor compliance
Quality of life under anticoagulants evaluation by Anti-Clot Treatment Scale (ACTS) satisfaction scores between the 2 arms | From enrollment to the end of follow-up (24 months post-inclusion or thrombotic recurrence)
  Anti-Clot Treatment Scale (ACTS) satisfaction scores measured at inclusion and at follow-up visits.
  The ACTS Burdens total score ranges from 12 to 60, and the ACTS Benefits total score ranges from 3 to 15. A high score for both indicates better quality of life on anticoagulants

CONTACTS AND LOCATIONS:
Overall Officials: Virginie DUFROST, MD, Principal Investigator — CHRU - Nancy
Locations (13):
- France (13):
  - Central Hospital, Nancy, France, Vandœuvre-lès-Nancy, Grand Est
  - CHU d'Amiens, Amiens
  - CHU de Besançon, Besançon
  - CHU de Brest, Brest
  - CHU de Dijon, Dijon
  - CHU de Lyon, Lyon
  - Hôpital Robert Schuman, UNEOS, Metz
  - CH de Mulhouse, Mulhouse
  - CHU de Nantes, Nantes
  - Hôpital Lariboisière - APHP, Paris
  - CHU de Reims, Reims
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - CHU de Strasbourg - Hôpital civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams B, Saseen JJ, Trujillo T, Palkimas S. Direct oral anticoagulants versus warfarin in patients with single or double antibody-positive antiphospholipid syndrome. J Thromb Thrombolysis. 2022 Jul;54(1):67-73. doi: 10.1007/s11239-021-02587-0. Epub 2021 Nov 24. PMID 34817786
- [Background] Dufrost V, Darnige L, Reshetnyak T, Vorobyeva M, Jiang X, Yan XX, Gerotziafas G, Jing ZC, Elalamy I, Wahl D, Zuily S. New Insights into the Use of Direct Oral Anticoagulants in Non-high Risk Thrombotic APS Patients: Literature Review and Subgroup Analysis from a Meta-analysis. Curr Rheumatol Rep. 2020 May 20;22(7):25. doi: 10.1007/s11926-020-00901-y. PMID 32436109
- [Background] Zuily S, Cohen H, Isenberg D, Woller SC, Crowther M, Dufrost V, Wahl D, Dore CJ, Cuker A, Carrier M, Pengo V, Devreese KMJ. Use of direct oral anticoagulants in patients with thrombotic antiphospholipid syndrome: Guidance from the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. J Thromb Haemost. 2020 Sep;18(9):2126-2137. doi: 10.1111/jth.14935. PMID 32881337
- [Background] Dufrost V, Risse J, Reshetnyak T, Satybaldyeva M, Du Y, Yan XX, Salta S, Gerotziafas G, Jing ZC, Elalamy I, Wahl D, Zuily S. Increased risk of thrombosis in antiphospholipid syndrome patients treated with direct oral anticoagulants. Results from an international patient-level data meta-analysis. Autoimmun Rev. 2018 Oct;17(10):1011-1021. doi: 10.1016/j.autrev.2018.04.009. Epub 2018 Aug 11. PMID 30103045
- [Background] Pengo V, Denas G, Zoppellaro G, Jose SP, Hoxha A, Ruffatti A, Andreoli L, Tincani A, Cenci C, Prisco D, Fierro T, Gresele P, Cafolla A, De Micheli V, Ghirarduzzi A, Tosetto A, Falanga A, Martinelli I, Testa S, Barcellona D, Gerosa M, Banzato A. Rivaroxaban vs warfarin in high-risk patients with antiphospholipid syndrome. Blood. 2018 Sep 27;132(13):1365-1371. doi: 10.1182/blood-2018-04-848333. Epub 2018 Jul 12. PMID 30002145